CLINICAL TRIAL: NCT01034254
Title: Field Trial of Maternal Influenza Immunization in Asia
Acronym: Mothers'Gift
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Seattle Children's Hospital (Other); Tribhuvan University, Nepal (Other); Johns Hopkins Bloomberg School of Public Health (Other); Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Mothers'Gift 241 Field Trial
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Influenza Human
Keywords: influenza; immunization; pregnancy; efficacy; pertussis; hepatitis E
MeSH Terms: conditions — Influenza, Human; Whooping Cough; Hepatitis E | interventions — Influenza Vaccines; vaxigrip; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- influenza vaccine (Experimental): Pregnant women assigned to the intervention group will receive one dose of seasonal influenza vaccine at the time of enrollment. The vaccine that will be given will be the current seasonal influenza recommended vaccine at the time of enrollment.
  Interventions: Biological: influenza vaccine
- saline placebo (Placebo Comparator): Pregnant women assigned to the control group will receive one dose of placebo (normal saline).
  Interventions: Biological: saline placebo

INTERVENTIONS:
Biological: influenza vaccine — Pregnant women will receive FDA approved influenza vaccine.
  Other Names: "VAXIGRIP®
  Arms: influenza vaccine
Biological: saline placebo — Vaccination of pregnant women with saline placebo.
  Other Names: saline
  Arms: saline placebo

SUMMARY:
This project is designed to assess the efficacy of immunizing women during pregnancy with influenza vaccine on the health of these women during their pregnancy and for 6 months post-partum as well as on the health of their newborn infants during the first 6 months of life. It will be conducted in Sarlahi District in southern Nepal, a rural area where a number of large scale randomized trials have been conducted over the past 20 years.

DETAILED DESCRIPTION:
This is a community-based, placebo-controlled, individually randomized trial in trial among women who are or who become pregnant in 9 Village Development Committees in Sarlahi District, Nepal. The study population for this trial will include all women who are identified as pregnant with gestational age between 17 and 34 weeks gestation during a 12-month period in 9 Village Development Committees (VDC) of Sarlahi District, Nepal. The 9 VDCs include: Dhungre Khola, Karmaiya, Hariaun, Ghurkauli, Sasapur, Netraganj, Lalbandi, Jabdi, and Raniganj.

The vaccine that will be given will be the most current vaccine at the time of subject enrollment. That is, for women enrolled after October in either study cohort, the vaccine will be switched to the newly available vaccine for that year.

The control group will be placebo (saline injection). The justification for the use of a placebo injection in this trial is as follows: There is only one trial (Bangladesh) that demonstrates efficacy of influenza vaccination in pregnancy on perinatal outcomes and respiratory morbidity in early infancy. One of the issues with that study is that it was not placebo controlled. The "control" in that study was adult pneumococcal vaccine. It could be that the Bangladesh study underestimated the impact of influenza vaccine because the mothers and infants receive some indirect protection from the pneumococcal vaccine. In addition, influenza vaccine is not part of national policy or recommendations in Nepal at the current time and Ministry of Health officials are very interested in the results of our study as they consider their immunization program expansion over the next few years.

ELIGIBILITY:
Inclusion Criteria:

* mid to late pregnancy

Exclusion Criteria:

* do not intend to deliver in the study area
* previous pregnancy in this study

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3693 (Actual)
Dates: Start 2010-11; Primary Completion 2014-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Field Trial of Maternal Influenza Immunization | 2 annual recruitment cycles coinciding with flu seasons
  To compare, in women randomized to receive either influenza vaccine or control during pregnancy and their infants (through 6 months of age)
  a) the incidence of influenza-like illness or lab-confirmed influenza episodes b) the distribution of causes of febrile illness and the incidence of clinic visits and hospitalizations c) the incidence of low birth weight, the distribution of birth weight and gestational age and the growth of infants.

SECONDARY OUTCOMES:
Substudy #1: Transplacental Transfer of Influenza Antibody from Mother to Infant | 2 annual recruitment cycles
  1. To estimate the efficacy of maternal vaccination for producing an immune response in the mother and for passive antibody transfer to the infant.
  2. To determine if timing of vaccination during pregnancy or other maternal factors such as nutritional status are related to level of antibody transfer to the infant.
  3. To compare neutralizing antibody concentrations in breastmilk of women randomized to receive either influenza vaccine or control during pregnancy.
Substudy #2: Indirect Protection of Maternal Influenza Vaccination on Family Members | 2 annual recruiting cycles
  Specific Aim: To compare the indirect protection of influenza vaccine on influenza-like and influenza-specific febrile illness rates in families of study women.
Substudy #3: Hepatitis E Infection in Pregnancy | 2 annual recruiting cycles
  1. To estimate the prevalence of anti-hepatitis E immunoglobulin G in women of reproductive age in rural Nepal.
  2. To estimate the incidence of hepatitis E infection (anti-hepatitis E seroconversion) during pregnancy in rural Nepal.
     1. To estimate the disease to infection ratio among women who seroconvert.
     2. To evaluate biochemical correlates of clinical disease among women who seroconvert.
  3. To describe pregnancy outcomes (miscarriage, stillbirth, neonatal mortality, maternal mortality) associated with women identified with incident infection or acute hepatitis E disease.
Pertussis In Infants | 2 annual rucruiting cycles
  Estimate the incidence of pertussis in infants under 6 months of age and the protection afforded by maternal antibody transfer to infants.

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Steinhoff, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Institute of Medicine, Tribhuvan Univerisity, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Undecided
To be determined

REFERENCES:
- [Background] Cox S, Posner SF, McPheeters M, Jamieson DJ, Kourtis AP, Meikle S. Hospitalizations with respiratory illness among pregnant women during influenza season. Obstet Gynecol. 2006 Jun;107(6):1315-22. doi: 10.1097/01.AOG.0000218702.92005.bb. PMID 16738158
- [Background] Dodds L, McNeil SA, Fell DB, Allen VM, Coombs A, Scott J, MacDonald N. Impact of influenza exposure on rates of hospital admissions and physician visits because of respiratory illness among pregnant women. CMAJ. 2007 Feb 13;176(4):463-8. doi: 10.1503/cmaj.061435. PMID 17296958
- [Background] Englund JA. Maternal immunization with inactivated influenza vaccine: rationale and experience. Vaccine. 2003 Jul 28;21(24):3460-4. doi: 10.1016/s0264-410x(03)00351-7. PMID 12850360
- [Background] Greenwood B. Maternal immunisation in developing countries. Vaccine. 2003 Jul 28;21(24):3436-41. doi: 10.1016/s0264-410x(03)00346-3. PMID 12850355
- [Background] Healy CM, Baker CJ. Maternal immunization. Pediatr Infect Dis J. 2007 Oct;26(10):945-8. doi: 10.1097/INF.0b013e318156c18c. No abstract available. PMID 17901801
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534
- [Background] Mak TK, Mangtani P, Leese J, Watson JM, Pfeifer D. Influenza vaccination in pregnancy: current evidence and selected national policies. Lancet Infect Dis. 2008 Jan;8(1):44-52. doi: 10.1016/S1473-3099(07)70311-0. PMID 18156088
- [Background] Zaman K, Roy E, Arifeen SE, Rahman M, Raqib R, Wilson E, Omer SB, Shahid NS, Breiman RF, Steinhoff MC. Effectiveness of maternal influenza immunization in mothers and infants. N Engl J Med. 2008 Oct 9;359(15):1555-64. doi: 10.1056/NEJMoa0708630. Epub 2008 Sep 17. PMID 18799552
- [Background] MacDonald NE, Riley LE, Steinhoff MC. Influenza immunization in pregnancy. Obstet Gynecol. 2009 Aug;114(2 Pt 1):365-368. doi: 10.1097/AOG.0b013e3181af6ce8. PMID 19622998
- [Background] Tamma PD, Ault KA, del Rio C, Steinhoff MC, Halsey NA, Omer SB. Safety of influenza vaccination during pregnancy. Am J Obstet Gynecol. 2009 Dec;201(6):547-52. doi: 10.1016/j.ajog.2009.09.034. Epub 2009 Oct 21. PMID 19850275
- [Background] Pickering LK, Baker CJ, Freed GL, Gall SA, Grogg SE, Poland GA, Rodewald LE, Schaffner W, Stinchfield P, Tan L, Zimmerman RK, Orenstein WA; Infectious Diseases Society of America. Immunization programs for infants, children, adolescents, and adults: clinical practice guidelines by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Sep 15;49(6):817-40. doi: 10.1086/605430. PMID 19659433
- [Background] Fiore AE, Shay DK, Broder K, Iskander JK, Uyeki TM, Mootrey G, Bresee JS, Cox NS; Centers for Disease Control and Prevention (CDC); Advisory Committee on Immunization Practices (ACIP). Prevention and control of influenza: recommendations of the Advisory Committee on Immunization Practices (ACIP), 2008. MMWR Recomm Rep. 2008 Aug 8;57(RR-7):1-60. PMID 18685555
- [Derived] Regodon Wallin A, Tielsch JM, Khatry SK, Mullany LC, Englund JA, Chu H, LeClerq SC, Katz J. Nausea, vomiting and poor appetite during pregnancy and adverse birth outcomes in rural Nepal: an observational cohort study. BMC Pregnancy Childbirth. 2020 Sep 17;20(1):545. doi: 10.1186/s12884-020-03141-1. PMID 32943001
- [Derived] Omer SB, Clark DR, Madhi SA, Tapia MD, Nunes MC, Cutland CL, Simoes EAF, Aqil AR, Katz J, Tielsch JM, Steinhoff MC, Wairagkar N; BMGF Supported Maternal Influenza Immunization Trials Investigators Group. Efficacy, duration of protection, birth outcomes, and infant growth associated with influenza vaccination in pregnancy: a pooled analysis of three randomised controlled trials. Lancet Respir Med. 2020 Jun;8(6):597-608. doi: 10.1016/S2213-2600(19)30479-5. PMID 32526188
- [Derived] Clark DR, Omer SB, Tapia MD, Nunes MC, Cutland CL, Tielsch JM, Wairagkar N, Madhi SA; for BMGF Supported Maternal Influenza Immunization Trials Investigators Group. Influenza or Meningococcal Immunization During Pregnancy and Mortality in Women and Infants: A Pooled Analysis of Randomized Controlled Trials. Pediatr Infect Dis J. 2020 Jul;39(7):641-644. doi: 10.1097/INF.0000000000002629. PMID 32379201
- [Derived] Murray AF, Englund JA, Kuypers J, Tielsch JM, Katz J, Khatry SK, Leclerq SC, Chu HY. Infant Pneumococcal Carriage During Influenza, RSV, and hMPV Respiratory Illness Within a Maternal Influenza Immunization Trial. J Infect Dis. 2019 Aug 9;220(6):956-960. doi: 10.1093/infdis/jiz212. PMID 31056697
- [Derived] Katz J, Englund JA, Steinhoff MC, Khatry SK, Shrestha L, Kuypers J, Mullany LC, Chu HY, LeClerq SC, Kozuki N, Tielsch JM. Impact of Timing of Influenza Vaccination in Pregnancy on Transplacental Antibody Transfer, Influenza Incidence, and Birth Outcomes: A Randomized Trial in Rural Nepal. Clin Infect Dis. 2018 Jul 18;67(3):334-340. doi: 10.1093/cid/ciy090. PMID 29452372
- [Derived] Omer SB, Clark DR, Aqil AR, Tapia MD, Nunes MC, Kozuki N, Steinhoff MC, Madhi SA, Wairagkar N; for BMGF Supported Maternal Influenza Immunization Trials Investigators Group. Maternal Influenza Immunization and Prevention of Severe Clinical Pneumonia in Young Infants: Analysis of Randomized Controlled Trials Conducted in Nepal, Mali and South Africa. Pediatr Infect Dis J. 2018 May;37(5):436-440. doi: 10.1097/INF.0000000000001914. PMID 29443825
- [Derived] Katz J, Englund JA, Steinhoff MC, Khatry SK, Shrestha L, Kuypers J, Mullany LC, Chu HY, LeClerq SC, Kozuki N, Tielsch JM. Nutritional status of infants at six months of age following maternal influenza immunization: A randomized placebo-controlled trial in rural Nepal. Vaccine. 2017 Dec 4;35(48 Pt B):6743-6750. doi: 10.1016/j.vaccine.2017.09.095. Epub 2017 Oct 31. PMID 29100709
- [Derived] Kozuki N, Katz J, Englund JA, Steinhoff MC, Khatry SK, Shrestha L, Kuypers J, Mullany LC, Chu HY, LeClerq SC, Tielsch JM. Impact of maternal vaccination timing and influenza virus circulation on birth outcomes in rural Nepal. Int J Gynaecol Obstet. 2018 Jan;140(1):65-72. doi: 10.1002/ijgo.12341. Epub 2017 Nov 9. PMID 28984909
- [Derived] Steinhoff MC, Katz J, Englund JA, Khatry SK, Shrestha L, Kuypers J, Stewart L, Mullany LC, Chu HY, LeClerq SC, Kozuki N, McNeal M, Reedy AM, Tielsch JM. Year-round influenza immunisation during pregnancy in Nepal: a phase 4, randomised, placebo-controlled trial. Lancet Infect Dis. 2017 Sep;17(9):981-989. doi: 10.1016/S1473-3099(17)30252-9. Epub 2017 May 15. PMID 28522338
- [Derived] Tielsch JM, Steinhoff M, Katz J, Englund JA, Kuypers J, Khatry SK, Shrestha L, LeClerq SC. Designs of two randomized, community-based trials to assess the impact of influenza immunization during pregnancy on respiratory illness among pregnant women and their infants and reproductive outcomes in rural Nepal. BMC Pregnancy Childbirth. 2015 Feb 20;15:40. doi: 10.1186/s12884-015-0470-y. PMID 25879974